CLINICAL TRIAL: NCT00884728
Title: East Arnhem Healthy Skin Project: A Regional Collaboration to Reduce Scabies, Skin Sores and Associated Chronic Diseases, Including Rheumatic Fever and Renal Disease, Among Australian Aboriginal Communities
Brief Title: Evaluation of a Regional Healthy Skin Program in Remote Aboriginal Communities of Australia's Northern Territory
Acronym: EAHSP
Status: Completed | Type: Observational
Sponsor: Menzies School of Health Research (Other)
Collaborators: University of Melbourne (Other); Murdoch Childrens Research Institute (Other); Cooperative Research Centre for Aboriginal Health (Other)
Responsible Party: Professor Jonathan Carapetis, Menzies School of Health Research
Other Study IDs: 41 17May2004
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Scabies; Impetigo; Pyoderma; Streptococcal Infections
Keywords: Scabies; Impetigo; Pyoderma; Streptococcal infections
MeSH Terms: conditions — Scabies; Impetigo; Pyoderma; Streptococcal Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — throat swabs, pyoderma swabs and skin scrapings for tinea where individual consent was obtained within selected participating communities
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Indigenous children aged <15 years: Indigenous children aged <15 years within participating communities of the Northern Territory

SUMMARY:
The purpose of this study is to determine whether a coordinated regional approach to healthy skin programs in six remote Aboriginal communities can demonstrate, not only a reduction in the burden of scabies and streptococcal skin sores, but also broad health benefits, including primary prevention of some chronic diseases that occur at particularly high rates in Australian Aboriginal communities.

The primary objectives of the Program are:

* Demonstrate a reduction in scabies and skin sores on a regional basis
* Demonstrate the broader public health effects of Healthy Skin Programs, particularly those relating to chronic diseases such as rheumatic fever and renal diseases
* Build on the existing Indigenous capacity by assisting in the development of new knowledge and skills to improve the health and well being of Indigenous communities
* Establish the feasibility of incorporating Healthy Skin Programs into existing health service delivery

DETAILED DESCRIPTION:
There are standard government recommendations for the conduct of healthy skin programs within the Northern Territory (NT), where the key component involves a single mass treatment for scabies of all residents in the region followed by regular monitoring of skin infections with treatment of individuals as new cases arise. The key features of the guidelines include:

* Community planning and collaborative effort;
* Development of local educational resources;
* Single whole community treatment day for scabies with permethrin (5%);
* Community "clean up" involving house cleaning, linen and rubbish collection;
* Emphasis on housing functionality and "washing kids" to maintain low rates of skin sores; and
* Regular monitoring of scabies and skin sores, usually in a target group such as children

Previous programs have been successful in controlling scabies and related skin infections in the NT but have been limited to single communities with varying levels of success. In collaboration with communities in the East Arnhem Region, we propose to conduct a coordinated Healthy Skin Program. By concentrating on one region, the project has an increased likelihood of success because reinfection due to mobility between communities will be minimised, and because the project will be recognised as a collaboration between multiple communities.

The program is structured into three distinct components:

* Implementation of the program within the participating communities;
* Evaluation of the program against specific outcomes; and
* Integration of the program into routine service delivery.

ELIGIBILITY:
Inclusion Criteria:

* All children aged <15 years in the participating communities

Exclusion Criteria:

* None

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Residents aged <15 years of participating communities in a remote region of the Northern Territory
Sampling Method: Non-Probability Sample
Enrollment: 2329 (Actual)
Dates: Start 2004-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Reduced prevalence of scabies among children in the participating communities from 30% (expected prevalence pre-program) to <10% at least 2 years following the introduction of the program | 2 years
Reduced prevalence of skin sores among children in the participating communities from 50% (expected prevalence pre-program) to <25% at least 2 years following the introduction of the program | 2 years

SECONDARY OUTCOMES:
Reduced severity of skin sores among children in the participating communities from 40% classified as moderate/severe (expected pre-program) to <15% classified as moderate/severe at least two years following the introduction of the program | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ross M Andrews, PhD, Principal Investigator — Menzies School of Health Research; Jonathan R Carapetis, PhD, MBBS, Principal Investigator — Menzies School of Health Research; Bart Currie, MBBS, DTM&H, Principal Investigator — Menzies School of Health Research; Christine Connors, MBBS, Principal Investigator — Northern Territory Govermnent Department of Health and Families; Shelley Walton, PhD, Principal Investigator — Menzies School of Health Research; Colin J Parker, MBBS, Principal Investigator — Australasian College of Dermatologists
Locations (1):
- Menzies School of Health Research, Casuarina, Northern Territory, Australia

REFERENCES:
- [Derived] Andrews RM, Kearns T, Connors C, Parker C, Carville K, Currie BJ, Carapetis JR. A regional initiative to reduce skin infections amongst aboriginal children living in remote communities of the Northern Territory, Australia. PLoS Negl Trop Dis. 2009 Nov 24;3(11):e554. doi: 10.1371/journal.pntd.0000554. PMID 19936297